CLINICAL TRIAL: NCT02612571
Title: Comparing Rates of Glaucomatous Optic Neuropathy in Professional Wind Versus Non-wind Instrument Players in the Philadelphia Orchestra
Brief Title: Comparing Rates of Glaucoma in Professional Wind Versus Non-Wind Instrument Players
Status: Completed | Type: Observational
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, L. Jay Katz MD, Principal Investigator, Wills Eye
Other Study IDs: 15-495
Record Dates: First submitted 2015-08-06; First posted 2015-11-24 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Glaucoma; Intraocular Pressure; Optic Neuropathy
MeSH Terms: conditions — Glaucoma; Optic Nerve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Wind instrument players: A wind instrument is defined as any instrument that contains a resonator, in which a column of air is set into resonation by the player blowing into a mouthpiece at one end of the resonator.
- Non-wind instrument players: A non-wind instrument is defined as any instrument that does not contain a resonator.

SUMMARY:
The purpose of the present study is to compare rates of glaucomatous optic neuropathy in professional wind versus non-wind instrument players in the Philadelphia Orchestra. A secondary objective is to evaluate intra-ocular pressure and choroidal thickness of wind instrument players under variable playing conditions.

DETAILED DESCRIPTION:
Participants of this study will be any current or retired member of the Philadelphia Orchestra. Approximately 100 participants will be divided into 2 groups: 1) wind instrument players and 2) non-wind instrument players.

A wind instrument is defined as any instrument that contains a resonator, in which a column of air is set into resonation by the player blowing into a mouthpiece at one end of the resonator. A non-wind instrument is defined as any instrument that does not meet the wind instrument criteria.

On the day of the eye examinations, the investigator will provide a brief overview to explain the purpose and goals of the study to all potential participants. The examination team will be set up in an adjoining room. Members of the orchestra will be able to visit the examination team at any time during their practice session. A trained technician will perform the following for both eyes for all participants:visual acuity,undilated fundus color photography and intra-ocular pressure measurement. The investigators will record the examination findings using a standard form. Demographic information, including ocular, medical, social, and family history, will be documented for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Play wind or non-wind instrument for average of 1 hour per day for minimum of 5 years.
* Normal general health.

Exclusion Criteria:

* Incisional eye surgery <1 month prior to visit 1.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Current and retired members of the Philadelphia Orchestra who play or played wind and non-wind instruments for an average of 1 hour per day for a minimum of 5 years.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) in wind and non-wind instrument players | 1 year
  Compare IOP in wind and non-wind instrument players

CONTACTS AND LOCATIONS:
Overall Officials: L J Katz, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Manuscript has been written and submitted to American Journal of Ophthalmology.